CLINICAL TRIAL: NCT02221310
Title: A Pilot Study of Gemtuzumab Ozogamicin in Combination With Busulfan and Cyclophosphamide (Immunochemotherapy) and Allogeneic Stem Cell Transplantation in Patients With High Risk Acute Myelogenous Leukemia and Myelodysplastic Syndrome
Brief Title: Immunochemotherapy and AlloSCT in Patients With High Risk CD33+ AML/MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-515; L-10,349 (Other: New York Medical College)
Record Dates: First submitted 2014-07-31; First posted 2014-08-20 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: targeted therapy; leukemia; MDS; immune therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemtuzumab Ozogamicin (Experimental): Conditioning therapy with Gemtuzumab Ozogamicin in combination with busulfan and cyclophosphamide chemotherapy followed by allogeneic stem cell transplantation.
  Interventions: Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Gemtuzumab Ozogamicin 7.5 mg/m^2/dose given IV over 2 hours once during conditioning
  Other Names: Mylotarg

SUMMARY:
Targeted immune therapy with gemtuzumab ozogamicin (Mylotarg) in combination with chemotherapy followed by allogeneic stem cell transplantation will be given to patients with high risk acute myelogenous leukemia (AML) or myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
Gemtuzumab ozogamicin in combination with busulfan and cyclophosphamide (immunochemotherapy) conditioning followed by allogeneic stem cell transplantation + anti-thymocyte globulin (unrelated donors only) in patients with high risk CD33+AML or MDS meeting eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Disease Status:

  * History of AML Induction/Reinduction Failure
  * AML 1st Complete Remission (CR) with poor cytogenetics
  * AML 2nd CR with minimal residual disease (MRD)
  * AML 3rd CR
  * AML in refractory relapse but ≤25% bone marrow leukemia blasts
  * MDS with >6% bone marrow blasts at diagnosis
  * Secondary MDS with ≤5% bone marrow myeloblasts at diagnosis

Disease Immunophenotype:

• Disease must express a minimum of >/= 10% CD33+ for patients with AML

Organ Function:

• Adequate renal function, adequate liver function, adequate cardiac function, adequate pulmonary function Age: ≤25 years of age Donor: matched family donor, unrelated cord blood donor, unrelated adult donor

Exclusion Criteria:

* Patients with active central nervous system (CNS) AML/MDS disease at time of conditioning therapy
* Female patients who are pregnant
* Karnofsky <50% or Lansky <50% if 10 years or less
* Age >25 years
* Has received gemtuzumab in the previous 30 days or has not recovered from prior gemtuzumab therapy.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-12-07 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 year
  overall response rate (CR + PR) in patients receiving GO, busulfan and cyclophosphamide and AlloSCT in patients with measurable disease (relapse/refractory) with high risk CD33+ AML/MDS

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Satwani P, Bhatia M, Garvin JH Jr, George D, Dela Cruz F, Le Gall J, Jin Z, Schwartz J, Duffy D, van de Ven C, Foley S, Hawks R, Morris E, Baxter-Lowe LA, Cairo MS. A Phase I study of gemtuzumab ozogamicin (GO) in combination with busulfan and cyclophosphamide (Bu/Cy) and allogeneic stem cell transplantation in children with poor-risk CD33+ AML: a new targeted immunochemotherapy myeloablative conditioning (MAC) regimen. Biol Blood Marrow Transplant. 2012 Feb;18(2):324-9. doi: 10.1016/j.bbmt.2011.11.007. Epub 2011 Nov 9. PMID 22079471